CLINICAL TRIAL: NCT01749124
Title: "My Coach Connect": Pilot Under the Partnered Research Center for Quality Care, RHINO 2008-0132
Brief Title: My Coach Connect: An Automated Telephone-based Reporting System for Patients With Mental Illness
Acronym: MCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: RHINO 2008-0132; P30MH082760 (NIH)
Record Dates: First submitted 2012-12-11; First posted 2012-12-13 (Estimated); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Chronic Mental Illness; Major Depression; Schizophrenia; Bipolar Disorder
Keywords: mental illness; depression; schizophrenia; bipolar disorder; IVR; automated; telephone
MeSH Terms: conditions — Depressive Disorder, Major; Schizophrenia; Bipolar Disorder; Mental Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- My Coach Connect (Experimental): To evaluate the feasibility and effectiveness of this telephone tool while engaging clients and providers in discussion groups and surveys to better understand how this tool impacts the care provided and their overall experience in healthcare. Clients will use this tool to leave voice messages and survey answers which their providers will have access to by logging in to a secure website. Providers will have access to audio recordings of the voice responses, transcribed text of the responses, as well as "word clouds" generated from the text. Word clouds are a method of displaying the content of text such that words that are used more frequently are displayed in a larger size than words used less frequently.
  Interventions: Behavioral: My Coach Connect

INTERVENTIONS:
Behavioral: My Coach Connect — Clients will call in to the system approximately twice a week for a period of four months. The study will be conducted in two phases. There will be an initial pilot phase where we will seek to enroll approximately 15-20 patients and 2-3 providers. This phase will last approximately two months and the goal will be to assess feasibility and obtain feedback on the tool and surveys to optimize them for this setting. We will begin the main phase of the study approximately one month after the end of the first phase and in that study seek to recruit approximately 150 patients and 5-10 providers from the ROADS program. Clients enrolled in this main phase of the study will enroll for a period of four months.
  Other Names: MCC

SUMMARY:
This is a pilot study for a novel, automated telephone system called "My Coach Connect". The purpose of the study is to evaluate the feasibility and effectiveness of this telephone tool while engaging clients and providers in discussion groups and surveys to better understand how this tool impacts the care provided and their overall experience in healthcare.

DETAILED DESCRIPTION:
Clients will use this tool (My Coach Connect) to leave voice messages and survey answers which their providers will have access to by logging in to a secure website. Providers will also be able to indicate using the website whether they found a particular narrative helpful or not. Providers will have access to audio recordings of the voice responses, transcribed text of the responses, as well as "word clouds" generated from the text. Word clouds are a method of displaying the content of text such that words that are used more frequently are displayed in a larger size than words used less frequently. Clients will call in to the system approximately twice a week for a period of four months.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the ROADS program
* English speaking
* Have a working telephone

Exclusion Criteria:

* Must speak english

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2012-12-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Client and provider telephone intervention | four months
  Clients will call in to an automated telephone system twice a week and will answer open-ended questions related to how they are doing. In addition, the system will prompt them to complete an automated SF-12 survey every four weeks to assess their mental and physical health status. The content of the voice messages will be made available to the providers as described above. Providers will also be able to indicate using the website whether they found a particular narrative helpful or not. One of the goals of the study is to determine if there is a correlation between the content of the client's messages and their overall health status. To investigate this, we will combine the content of the voice messages with information obtained from the client's medical record including provider observations, assessment, and symptom recording.

SECONDARY OUTCOMES:
Client and provider survey | 4 months
  Each client and provider will be asked to complete a brief survey about their expectations, thoughts and experiences while participating in this study. The survey will be conducted at the time of enrollment as well as the time of disenrollment or completion of the study as a comparison.

OTHER OUTCOMES:
Discussion groups | 4 months
  To better understand the impact of the tool on participants that use it and how to improve the tool, we will also organize discussion groups that clients and providers will have the opportunity to participate in.

CONTACTS AND LOCATIONS:
Overall Officials: Ken Wells, MD, MPH, Principal Investigator — RAND; Armen Arevian, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- ROADS (Recovery, Opportunity, And Developing Skills), Long Beach, California, United States

IPD SHARING:
Plan to Share IPD: No